CLINICAL TRIAL: NCT04894370
Title: Spartalizumab, mDCF (Docetaxel, Cisplatin and 5-fluorouracil) and Radiotherapy in Patients With Metastatic Squamous Cell Anal Carcinoma. A Phase IIA Study
Brief Title: Combination of Spartalizumab, mDCF and Radiotherapy in Patients With Metastatic Squamous Cell Anal Carcinoma
Acronym: SPARTANA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: National Cancer Institute, France (Other Government); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/538
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Squamous Cell Anal Carcinoma; Metastatic Squamous Cell Carcinoma
Keywords: immunotherapy; chemotherapy; radiotherapy; anti-PD1
MeSH Terms: conditions — Anus Neoplasms; Carcinoma, Squamous Cell | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Phase 1: Radiotherapy (8 Gy on target lesions)
  Phase 2: Combination immunotherapy and mDCF regimen mDCF regimen every 2 weeks for 8 cycles
  * Docetaxel (40 mg/m², day 1),
  * Cisplatin (40 mg/m², day 1)
  * 5-FU (1200 mg/m²/day for 2 days) Spartalizumab: 400 mg intravenous will be administrated every 4 weeks
  Phase 3 : Multimodal treatment of residual disease The multimodal treatment is recommended in oligometastatic anal cancer. The support by ablative treatment (surgery, hypofractionnated radiotherapy or by radiofrequency) improve survival.
  In absence of progression disease:
  * Ablative treatment: surgery, hypofractionnated radiotherapy or by radiofrequency of residual metastases
  * and Chemo-radiotherapy (CRT) for local disease
  Phase 4: Maintenance treatment with Spartalizumab 400 mg intravenous every 4 weeks for 12 months from enrolment maximum
  Interventions: Biological: Sample collection

INTERVENTIONS:
Biological: Sample collection — PBMC collection at baseline, after radiotherapy 8 Gy (gray), at 6 months and at 12 months from inclusion: 6 EDTA tubes of 6 ml of peripheral blood mononuclear cell [PBMC] will be sent to the central laboratory (Biomonitoring Platform of Besançon, CHRU de Besançon located at Etablissement Français du Sang) at room temperature within 24 hours via an approved carrier for their processing, storage and immunomonitoring analysis. A sending sheet of the samples will be attached to each single sample.
  Plasma collection at baseline, after radiotherapy 8 Gy, at 6 months and at 12 months from inclusion: One 6 ml EDTA tube should be frozen in each investigation center for plasma collection.
  Plasma for circulating tumoral DNA (ctDNA) collection at baseline, at 2, 6 and 12 months from inclusion: two EDTA tube of 4 ml should be frozen in each investigation center for ctDNA collection.

SUMMARY:
This study evaluates the feasibility of the combination of radiotherapy, chemotherapies (docetaxel, cisplatin and 5-fluorouracil) and spartalizumab (anti-PD-1 therapy) in patients with metastatic squamous cell anal carcinoma

DETAILED DESCRIPTION:
In SCCA (squamous cell carcinoma of anus) about 15% of patients are diagnosed in metastatic stage, and around 25-40% of patients will experience disease progression after curative intent chemoradiotherapy (CRT) for localized disease. In patients with non-resectable local recurrences or with distant metastases, the systemic chemotherapy is the standard approach. Recently, taxane-based combination chemotherapy regimens have demonstrated high efficacy or better tolerance than non-taxane based regimens, and became standards based in prospective trials. First, the modified DCF (docetaxel, cisplatin and 5-fluorouracil) showed a high efficacy in Epitopes-HPV02 trial conducted by investigators including 66 patients and became the first validated chemotherapy regimen in advanced SCCA. Then, the pooled analysis of 115 patients confirmed the mDCF regimen as the standard treatment in all fit patients with advanced SCCA.

The combination of different chemotherapy regimens and an anti-PD1/PD-L1 (Programmed cell Death-1/Programmed cell Death-Ligand1) were feasible with improved survival in first-line advanced small-cell and non-small-cell lung cancers. In anal carcinoma, Epitopes-HPV02 trial showed that mDCF regimen was feasible with 53% of grade 3-4 adverse-event, with no grade 4 non-hematological toxicity and no febrile neutropenia. And also considering its property to enhance the anti-tumor immune response, mDCF was recommended as an interesting candidate to be evaluated as a backbone chemotherapy for immunotherapy combinations in SCCA.

In anal carcinoma, investigators are currently conducting a randomized prospective trial promoted by GERCOR (cooperator group) evaluating the association of mDCF and an anti-PD-L1 in metastatic setting. All patients (100) were already enrolled, and no particular safety alert signal was observed at the Data Safety Monitoring Board (DSMB)..

Among different factors that confers a primary resistance to immunotherapy, the lack of antigenic proteins capable to induce immune response, and the downregulation of major histocompatibility complex class 1 (MHC-1) are probably the most important. In fact, the next-generation sequencing (NGS) techniques has demonstrated the correlation between tumor mutation burden (TMB) and response to CKI (checkpoint Inhibitor). Hence, most of "hot" tumors with high TMB could be treated with CKI alone, while "cold" tumors probably need combination strategies. Besides, primary or secondary resistances to CKI caused by downregulation of MHC-1 are well described.

Radiation causes random point mutations and double-stranded breaks in the DNA and modulates the peptide repertoire, increasing tumour-related antigens and TMB to enhance anti-tumour immunity. Radiotherapy has also demonstrated to enhances MHC class I expression.

Investigators decided to associate radiotherapy, PD-1 (Programmed cell Death-1) inhibitor and mDCF (docetaxel, cisplatin and 5-fluorouracil) chemotherapy regimen to improve the efficacy with higher rate of long-lasting progression-free survivors and complete remissions. In addition, the associated extensive ancillary biomarker studies in tissues and peripheral blood will provide a unique opportunity to find out the potential synergic effect mechanism between mDCF, CKI and radiotherapy, as well as to improve our knowledge about underlying resistances.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years,
2. Performance status Eastern Cooperative Oncology Group World Health Organization (ECOG-WHO) ≤1,
3. Histologically proven metastatic or locally advanced recurrent squamous cell carcinoma of anus (SCCA)
4. Presence of a evaluable lesion on CT-scan/MRI assessed by RECIST v1.1 criteria,
5. Patient eligible to the mDCF regimen
6. CT scan performed within 30 days prior inclusion,
7. PET scan performed within 30 days prior inclusion
8. Life expectancy ≥12 months,
9. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   * Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L) without granulocyte colony-stimulating factor support.
   * White blood cell count ≥ 2500/mm3 (≥ 2.5 GI/L).
   * Platelets ≥ 100,000/mm3 (≥ 100 GI/L) without transfusion.
   * Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN), or ≤ 5 x ULN with documented liver metastases.
   * Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3 x ULN).
   * Serum albumin ≥ 2.8 g/dl.
   * Calculated creatinine clearance ≥ 60 mL/min (using the MDRD formula):
   * Urine protein/creatinine ratio (UPCR) ≤ 1 g/g
10. Signed and dated informed consent, to participate indicating that the subject has understood the purpose and the procedures required by the study and that he agrees to participate in the study and to comply with the requirements and restrictions inherent in this study
11. Patient affiliated to or beneficiary of French social security system
12. Ability to comply with the study protocol, in the Investigator's judgment

Exclusion Criteria:

1. HIV positive patient , CD4 count < 400 cells/mm3 (HIV test mandatory before inclusion)
2. Diagnosis of additional malignancy within 2 years prior to the inclusion with the exception for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy,
3. Any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study,
4. Current participation in a study of an investigational agent or in the period of exclusion,
5. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment,
6. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible,
7. Pregnancy, breast-feeding or absence/refusal of adequate contraception for fertile patients during the period of treatment and for 6 months from the last treatment administration,
8. Patient under guardianship, curatorship or under the protection of justice.
9. Inability to perform radiotherapy
10. Untreated or symptomatic central nervous system (CNS) lesion. However, patients are eligible if: a) all known CNS lesions have been treated with radiotherapy or surgery and b) patient remained without evidence of CNS disease progression ≥ 4 weeks after treatment and c) patients must be off corticosteroid therapy for ≥ 2 weeks
11. Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GMCSF, M-CSF), thrombopoietin mimetics or erythroid stimulating agents ≤ 2 weeks prior start of study treatment. If erythroid stimulating agents were initiated more than 2 weeks prior to the first dose of study treatment and the patient is on a stable dose, they can be maintained.
12. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment
13. Elevated Cardiac troponin T (cTnT) or cardiac troponin I (cTnI) elevation > 2x ULN
14. Systemic chronic steroid therapy (> 10mg/day prednisone or equivalent) or any immunosuppressive therapy 7 days prior to planned date of first dose of study treatment.

    Note: Topical, inhaled, nasal and ophthalmic steroids are allowed. For patients with adrenal insufficiency, replacement dose of prednisone > 10 mg/ day or equivalent are permitted
15. Active, known or suspected autoimmune disease or a documented history of autoimmune disease Note: Patients with vitiligo, controlled type I diabetes mellitus on stable insulin dose, residual autoimmune-related hypothyroidism only requiring hormone replacement or psoriasis not requiring systemic treatment are permitted.
16. Allogenic bone marrow or solid organ transplant
17. History of severe hypersensitivity reactions to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction
18. Pre-existing neuropathy, hearing problem, or cardiorespiratory pathology, which prevent the administration of cisplatin.
19. clinically significant active heart disease or myocardial infarction within 6 months
20. recent or concomitant treatment with brivudine
21. persistent toxicities related to prior treatment of grade greater than 1
22. History or current interstitial lung disease or non-infectious pneumonitis
23. History of major surgery within 28 days before treatment
24. Active infection
25. Active Hepatitis B infection (HBsAg positive)
26. Active hepatitis C (HCV RNA positive)
27. Pregnant or nursing (lactating) women confirmed by a positive hCG laboratory test within 72 hours prior to initiating study treatment.

    Note: Low levels of hCG may also be considered a tumor marker, therefore if low hCG levels are detected, another blood sample at least 4 days later must be taken to assess the kinetics of the increase and transvaginal ultrasound must be performed to rule out pregnancy.
28. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 7.5 months after stopping treatment with Spartalizumab.
29. Complete or partial deficit in dihydropyrimidine dehydrogenase (DPD) activity
30. Active inflammatory bowel disease Note: In case of a history of inflammatory bowel disease, it is advisable to take the advice of the referring gastroenterologist of the patient to ensure the absence of the evolution of inflammatory bowel disease (inflammatory thrust in progress) before the initiation of docetaxel treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) rate at 1 year. | 12 months from enrollment
  PFS rate at 1 year is defined as the number of patients alive without progression at 1 year divided by the overall number of patients evaluable for PFS status at 1 year.
  A patient is evaluable for PFS status at 1 year if he dies during the 1 year of follow up or if he is alive with a RECIST evaluation available at 1 year.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 12 months from enrollment
  Addition of complete response (CR) and partial response (PR) rates.
Overall survival (OS) | through study completion, an average of 3 years
  Delay from the date of inclusion to death from any cause , or the date of the last follow-up, at which point data will be censored
Progression-Free Survival (PFS) median. | through study completion, an average of 3 years
  Delay from the date of inclusion to the disease progression or death from any cause, whichever occurs first , or the date of the last follow-up, at which point data will be censored

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Georges-François Leclerc (CGFL), Dijon
  - Hôpital Franco-Britannique, Levallois-Perret
  - Centre Léon Bérard, Lyon
  - Hôpital Nord Franche Comté, Montbéliard

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim S, Francois E, Andre T, Samalin E, Jary M, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, De La Fouchardiere C, Smith D, Deberne M, Spehner L, Badet N, Adotevi O, Anota A, Meurisse A, Vernerey D, Taieb J, Vendrely V, Buecher B, Borg C. Docetaxel, cisplatin, and fluorouracil chemotherapy for metastatic or unresectable locally recurrent anal squamous cell carcinoma (Epitopes-HPV02): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2018 Aug;19(8):1094-1106. doi: 10.1016/S1470-2045(18)30321-8. Epub 2018 Jul 2. PMID 30042063
- [Background] Kim S, Meurisse A, Spehner L, Stouvenot M, Francois E, Buecher B, Andre T, Samalin E, Jary M, Nguyen T, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, de la Fouchardiere C, Boulbair F, Lakkis Z, Klajer E, Jacquin M, Taieb J, Vendrely V, Vernerey D, Borg C. Pooled analysis of 115 patients from updated data of Epitopes-HPV01 and Epitopes-HPV02 studies in first-line advanced anal squamous cell carcinoma. Ther Adv Med Oncol. 2020 Dec 4;12:1758835920975356. doi: 10.1177/1758835920975356. eCollection 2020. PMID 33329760
- [Background] Kim S, Buecher B, Andre T, Jary M, Bidard FC, Ghiringhelli F, Francois E, Taieb J, Smith D, de la Fouchardiere C, Desrame J, Samalin E, Parzy A, Baba-Hamed N, Bouche O, Tougeron D, Dahan L, El Hajbi F, Jacquin M, Rebucci-Peixoto M, Spehner L, Vendrely V, Vernerey D, Borg C. Atezolizumab plus modified docetaxel-cisplatin-5-fluorouracil (mDCF) regimen versus mDCF in patients with metastatic or unresectable locally advanced recurrent anal squamous cell carcinoma: a randomized, non-comparative phase II SCARCE GERCOR trial. BMC Cancer. 2020 Apr 25;20(1):352. doi: 10.1186/s12885-020-06841-1. PMID 32334548